CLINICAL TRIAL: NCT07306897
Title: Risk Factors for Postoperative Pulmonary Complications After Major Abdominal Surgery in Patients Aged 65 Years and Older: A Retrospective Observational Study
Brief Title: Postoperative Pulmonary Complications in Elderly Patients Undergoing Major Abdominal Surgery
Acronym: PPC65MAS
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Timuroğlu, MD, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: PPC65-MAS-2024
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Postoperative Complications
MeSH Terms: conditions — Pneumonia; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with postoperative pulmonary complications (PPC +): Group 1 - Patients with postoperative pulmonary complications (PPC +):
  This group includes patients aged 65 years and older who underwent major abdominal surgery and developed one or more postoperative pulmonary complications, as defined by EPCO criteria
- Group 2: Patients without postoperative pulmonary complications (PPC -): Group 2 - Patients without postoperative pulmonary complications (PPC -):
  This group includes patients aged 65 years and older who underwent major abdominal surgery but did not develop any postoperative pulmonary complications.

SUMMARY:
This study aims to identify the risk factors associated with postoperative pulmonary complications (PPCs) in patients aged 65 years and older who undergo major abdominal surgery.

The study is designed as a retrospective observational analysis using data from patient records.

Understanding these risk factors may help clinicians improve perioperative care and reduce the risk of respiratory problems after surgery in elderly patients.

DETAILED DESCRIPTION:
This is a retrospective observational study. No follow-up was performed; all data were collected from existing patient records.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older.
* Patients who underwent major abdominal surgery at [Institution Name].
* Availability of complete perioperative and postoperative clinical records.
* Postoperative hospital stay of at least 24 hours.

Exclusion Criteria:

* Patients younger than 65 years.
* Patients undergoing minor or non-abdominal surgery.
* Incomplete or missing perioperative or postoperative medical records.
* Patients who underwent emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of patients aged 65 years and older who underwent major abdominal surgery. Only patients with complete perioperative and postoperative medical records were included. Patients were retrospectively classified into two groups based on the occurrence of postoperative pulmonary complications (PPCs) within the first 24 hours after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Pulmonary Complications | Within 1 day after surgery
  The primary outcome is the occurrence of one or more postoperative pulmonary complications (PPCs) in patients aged 65 years and older undergoing major abdominal surgery. PPCs include pneumonia, respiratory failure, or need for reintubation, as defined by the European Perioperative Clinical Outcome (EPCO) criteria. Data were collected retrospectively from patient records during the postoperative hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Timuroğlu, Principal Investigator — ankara oncology trainig and research hospital
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective observational study using existing patient medical records. Individual participant data (IPD) will not be publicly shared to protect patient confidentiality and comply with institutional and ethical regulations. Aggregate data may be shared upon reasonable request.